CLINICAL TRIAL: NCT01577056
Title: Effect of Fish Oil Supplementation on Postprandial Lipid Metabolism in Familial Hypercholesterolaemia
Brief Title: Postprandial Lipid Metabolism in Familial Hypercholesterolaemia:Effects of Fish Oils
Acronym: FIFH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Western Australia (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Dick C Chan, Assistant Professor, The University of Western Australia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1028883; NHMRC1028883 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Hypertriglyceridaemia; Familial Hypercholesterolaemia
Keywords: Familial hypercholesterolaemia; Postprandial dyslipidaemia; Fish oil treatment; Cardiovascular disease
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type II; Cardiovascular Diseases | interventions — Fish Oils; Omacor; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Active Comparator)
  Interventions: Dietary Supplement: Fish oil capsule
- Placebo (Placebo Comparator): FH subjects with standard treatment (statin treatment)
  Interventions: Drug: HMG Coenzyme reductase

INTERVENTIONS:
Dietary Supplement: Fish oil capsule — 4g Omega capsule for 12 weeks
  Other Names: Omacor
  Arms: Fish oil
Drug: HMG Coenzyme reductase — All FH subjects are on standard statin treatment during study period
  Other Names: Statin
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fish oil supplementation is effective in the treatment of abnormal fat metabolism in subjects with elevated cholesterolaemia.

DETAILED DESCRIPTION:
The use of statin therapy in familial hypercholesterolaemia (FH) is known to reduce cardiovascular risk and is a first line recommendation, however, there is considerable residual risk predicted by the presence of fasting and post-prandial hypertriglyceridaemia.

This study will examine the effect of oral n-3 fatty acid ethyl esters supplementation (4g/day, Omacor) on postprandial hypertriglyceridaemia and post-prandial arterial function when administrated to FH patients at increased risk of cardiovascular disease due to their residual fasting hypertriglyceridaemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FH (genetically defined LDL-receptor mutation or Dutch score >8) on statin treatment only
* Hypertriglyceridaemia on a random blood sample (triglycerides >1.5mml/L)

Exclusion Criteria:

* Subjects with diabetes mellitus
* major systemic illness or use of steroids or other lipid-regulating drugs (such as niacin, fibrate and colesevelam)
* patients on hypocaloric diets or LDL apheresis; anaemia, haemorrhage and pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Postprandial changes in triglyceride-rich lipoprotein concentrations | 12 weeks
  Incremental area-under-the-curve (AUC) for triglycerides, apoB-48 and retinyl palmitate

SECONDARY OUTCOMES:
Triglyceride-rich lipoprotein kinetics | 12 weeks
  Kinetic studies of apoB48 and apoB-100 kinetics

CONTACTS AND LOCATIONS:
Overall Officials: Dick Chan, Phd, Principal Investigator — The University of Western Australia
Locations (1):
- School of Medicine & Pharmacology,University of Western Australia, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Ying Q, Chan DC, Pang J, Croyal M, Blanchard V, Krempf M, Watts GF. Effect of omega-3 fatty acid ethyl esters on postprandial arterial elasticity in patients with familial hypercholesterolemia. Clin Nutr ESPEN. 2023 Jun;55:174-177. doi: 10.1016/j.clnesp.2023.03.012. Epub 2023 Mar 21. PMID 37202042
- [Derived] Chan DC, Pang J, Barrett PH, Sullivan DR, Mori TA, Burnett JR, van Bockxmeer FM, Watts GF. Effect of omega-3 fatty acid supplementation on arterial elasticity in patients with familial hypercholesterolaemia on statin therapy. Nutr Metab Cardiovasc Dis. 2016 Dec;26(12):1140-1145. doi: 10.1016/j.numecd.2016.07.012. Epub 2016 Aug 3. PMID 27614801
- [Derived] Chan DC, Pang J, Barrett PH, Sullivan DR, Burnett JR, van Bockxmeer FM, Watts GF. omega-3 Fatty Acid Ethyl Esters Diminish Postprandial Lipemia in Familial Hypercholesterolemia. J Clin Endocrinol Metab. 2016 Oct;101(10):3732-3739. doi: 10.1210/jc.2016-2217. Epub 2016 Aug 4. PMID 27490922